CLINICAL TRIAL: NCT01744548
Title: A Pilot Randomised Controlled Trial (RCT) Examining The Feasibility, Acceptability And Efficacy Of Transdiagnostic Cognitive Behavioural Therapy (tCBT) For Depression And Anxiety In Older People.
Brief Title: A Pilot Trial Of Transdiagnostic Cognitive Behavioural Therapy (tCBT) For Depression And Anxiety In Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Siobhan Commins, Trainee Clinical Psychologist, King's College London
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12/LO/1462
Record Dates: First submitted 2012-12-02; First posted 2012-12-06 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- tCBT treatment (Experimental): Participants randomised to the tCBT treatment arm will receive 12 individual, 1-hour tCBT sessions based upon Barlow et al.'s (2011) Unifed Protocol for emotional disorders (UP).
  Interventions: Behavioral: tCBT treatment
- 7-week delayed tCBT treatment (No Intervention): Participants randomised to the delayed-treatment arm will receive a brief telephone call and complete the Hospital Anxiety and Depression Scale (HADS) in order to monitor risk and symptom deterioration during the 7-week delayed treatment phase. They will also receive TAU (e.g. Community Mental Health Team appointments, case reviews, etc) during this time. At the end of 7 weeks, participants in the delayed-treatment arm will crossover into the treatment arm and receive the tCBT intervention. This arm will serve as a control condition in order to enable between-group comparisons.

INTERVENTIONS:
Behavioral: tCBT treatment — The UP comprises 4 main treatment components: 1) psychoeducation about emotions and behaviour; 2) changing misappraisals about probabilities and consequences of negative experiences; 3) preventing avoidance of negative emotion triggers; and 4) modifying emotion-driven behaviours (e.g. hypervigilance, withdrawal). The manualised tCBT intervention will be adapted in order to account for a United Kingdom (UK) audience (as the manual was developed in the United States) and older people (as the manual was developed for working-age people).
  Other Names: transdiagnostic Cognitive Behavioural Therapy (tCBT)
  Arms: tCBT treatment

SUMMARY:
This study aims to evaluate the feasibility, acceptability and efficacy of transdiagnostic Cognitive Behavioural Therapy (tCBT) in comparison to delayed-treatment for depression and anxiety in older people. CBT is a form of 'talking therapy' that has been recommended by the National Institute of Clinical Excellence for the treatment of mood disorders. While traditional disorder-specific CBT has been found to be effective at alleviating individual mood disorders, it may be less effective when multiple mood disorders are present (i.e. when there is psychological comorbidity). tCBT is a form of CBT that targets cognitive and behavioural processes common to a range of mood disorders. Consequently, it may be better placed to address comorbidity than traditional CBT, both in terms of clinical and cost-effectiveness.

There is growing evidence that tCBT has beneficial effects on both depression and anxiety in working-age people. However, the potential benefits of this approach have not yet been examined in older people (in whom psychological comorbidity is a frequent problem). Therefore, this study will aim to recruit 22 older people who are experiencing symptoms of depression and anxiety from community mental health teams within the South London and Maudsley National Health Service Trust. Participants will be randomly allocated to receive either tCBT plus treatment-as-usual (TAU) or 7-week delayed tCBT plus TAU. tCBT will be delivered on an individual basis in 12 sessions, each lasting 1 hour, over 14 weeks. It will be delivered in outpatient clinics or within the participants residence, depending on mobility issues. A number of outcome measures will be used to evaluate the feasibility, acceptability and efficacy of tCBT, including ratings on mood questionnaires, rates of dropout and reasons for dropout. Outcome measures will be collected before the tCBT intervention starts (week 0/baseline), midway through the intervention (after the 6th tCBT session/week 7), at the end of the intervention (after the final tCBT session/week 14) and at 7-week follow-up (week 21) .

The main hypotheses are:

i. It will be feasible to adapt and establish a tCBT intervention for older people with comorbid depressive and anxiety disorders.

ii. The tCBT intervention will be acceptable to older people with comorbid depressive and anxiety disorders.

iii. The tCBT intervention will significantly reduce depression and anxiety symptoms relative to a delayed-treatment control condition.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older;
* Primary diagnosis of mild to severe depression or anxiety, together with clinical symptoms of another mood disorder (e.g. anxiety or depression respectively), or a diagnosis of mixed anxiety and depressive disorder;
* Scores between 8 to 30 (mild to severe range) on the Hamilton Anxiety Rating Scale (HARS) or between 8 to 22 (mild to severe range) on the Hamilton Depression Rating Scale (HDRS) for the primary diagnosis;
* Fluent in English;
* Sufficient literacy skills and sensory abilities to cope with the demands of the psychological intervention (e.g reading handouts, completing questionnaires etc).

Exclusion Criteria:

* Current diagnosis of Post Traumatic Stress Disorder (PTSD) or Complicated Grief;
* Presence of a severe and enduring mental health disorder (e.g. Schizophrenia);
* Presence of a developmental intellectual disability or cognitive impairment (e.g. a score below 26 on the Mini Mental State Examination);
* Presence of a personality disorder;
* Presence of a severe sensory impairment;
* Presence of a neurodegenerative disease (e.g. dementia) or neurological condition (e.g stroke);
* Current alcohol/substance abuse or dependence;
* Current suicidal risk;
* Receiving concurrent psychotherapy;
* Receiving concurrent pharmacotherapy where stabilisation of dosages has not occurred (e.g. where pharmacotherapy has been introduced or changed less than 8-weeks prior to recruitment).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS). This will assess symptom change over time in order to evaluate the efficacy of the tCBT intervention. | The HADS will be completed on a weekly basis throughout the tCBT intervention (from week 0 to week 14) and once again at 7-week follow-up (week 21).
  Self-report questionnaire.
  The HADS will be used to measure changes in anxiety and depression symptoms on a weekly basis over the course of the tCBT intervention (from week 0 to week 14), and once again at 7-week follow-up (week 21) to establish whether any treatment gains have been maintained.
  For those participants allocated to the delayed-intervention arm of the trial the HADS will be also be completed each week during the 7-week delay period (week 0 to week 7) to monitor changes in symptoms and suicidal ideation. After the delay period these participants will crossover to the intervention arm and be evaluated accordingly (e.g. throughout the tCBT intervention; week 7 to week 21, and at 7-week follow-up; week 28).
Hamilton Anxiety Rating Scale (HARS). This will assess symptom change over time in order to evaluate the efficacy of the tCBT intervention. | The HARS will be completed before the tCBT intervention starts (week 0/7), mid-way through the intervention (week 7/14), after the final tCBT session (week 14/21), and at 7-week follow-up (week 21/28).
  This is a clinician-rated assessment, which will be completed by a blind outcome assessor.
Hamilton Depression Rating Scale (HDRS). This will assess symptom change over time in order to evaluate the efficacy of the tCBT intervention. | The HDRS will be completed before the tCBT intervention starts (week 0/7), mid-way through the intervention (week 7/14), after the final tCBT session (week 14/21), and at 7-week follow-up (week 21/28).
  This is a clinician-rated assessment, which will be completed by a blind outcome assessor.

SECONDARY OUTCOMES:
Clinical Outcomes of Routine Evaluation - 10 (CORE-10). This will assess symptom change over time in order to evaluate the efficacy of the tCBT intervention. | The CORE-10 will be completed before the tCBT intervention begins (week 0/7), after the final tCBT session (week 14/21), and at 7-week follow-up (week 21/28).
  Self-report questionnaire.
Discharge Satisfaction Questionnaire (DSQ) | After the final tCBT session (week 14/21)
  Self-report questionnaire

OTHER OUTCOMES:
Acceptability of tCBT | After the the final tCBT session (week 14/21)
  Acceptability will be evaluated using the DSQ and based on attrition rates due to dissatisfaction with the intervention.
Feasibility of tCBT | After the final tCBT session (week 14/21)
  The feasibility of the tCBT intervention will be assessed based on attrition rates due to practical reasons (e.g. difficulty in attending due to mobility issues or physical health problems, etc) and clinician-rated judgments of the intervention (e.g. ease of delivery, etc).

CONTACTS AND LOCATIONS:
Locations (1):
- South London and Maudsley NHS Trust, South London, London, United Kingdom